CLINICAL TRIAL: NCT00650455
Title: Clinical Protocol for a Multicenter, Double-Blind, Randomized, Placebo Controlled, Comparison of the Efficacy and Safety of Bextra® (Valdecoxib) 10 mg Once Daily and Naproxen 500 mg Twice Daily in Treating the Signs and Symptoms of Rheumatoid Arthritis (RA) in a Severe RA Population
Brief Title: Efficacy and Safety of Valdecoxib and Naproxen in Treating the Signs and Symptoms of Rheumatoid Arthritis (RA) in a Severe Rheumatoid Arthritis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3471018
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Last update posted 2008-07-21 (Estimated); Status verified 2008-07

CONDITIONS: Arthritis, Rheumatoid
Keywords: valdecoxib, severe rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — valdecoxib; Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 2 (Active Comparator)
  Interventions: Drug: naproxen
- Arm 3 (Placebo Comparator)
  Interventions: Drug: placebo
- Arm 1 (Active Comparator)
  Interventions: Drug: valdecoxib

INTERVENTIONS:
Drug: valdecoxib — valdecoxib 10 mg tablet once daily for 12 weeks
  Arms: Arm 1
Drug: naproxen — naproxen 500 mg capsule twice daily for 12 weeks
  Arms: Arm 2
Drug: placebo — placebo tablet every morning and capsule every evening for 12 weeks
  Arms: Arm 3

SUMMARY:
The objectives of the study were to evaluate the efficacy, safety, and tolerability of valdecoxib 10 mg once daily (QD) or naproxen 500 mg twice daily (BID) versus placebo, and to assess the efficacy of valdecoxib 10 mg QD versus naproxen 500 mg BID, in treating the signs and symptoms of rheumatoid arthritis (RA) in a severe Rheumatoid Arthritis population.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of severe rheumatoid arthritis (RA) for at least 6 months
* The Rheumatoid Arthritis must have been treated with a stable regimen including a non-steroidal anti-inflammatory drug (NSAID), as well as methotrexate for at least 12 weeks -OR- an NSAID (for at least 12 weeks plus a tumor necrosis factor inhibitor (i.e., adalimumab [Humira®] for a minimum of 5 doses on a regular schedule, etanercept [Enbrel®] for 6 weeks, infliximab (Remicade®) for 3 doses and currently on a stable regimen of infusions not more than every 8 weeks)

Exclusion Criteria:

* A diagnosis of any other inflammatory arthritis or a secondary, noninflammatory type of arthritis (eg, osteoarthritis (OA) or fibromyalgia) that, in the investigator's opinion, was symptomatic enough to interfere with the evaluation of the effect of valdecoxib on the patient's primary diagnosis of Rheumatoid Arthritis were excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 489 (Actual)
Dates: Start 2003-02; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
ACR-20 criteria responder | Week 12

SECONDARY OUTCOMES:
Patient's Global Assessment of Disease Activity | Screening, Baseline, Week 1, Week 6, and Week 12
Duration of morning stiffness | Screening, Baseline, Week 1, Week 6, and Week 12
Incidence and time to withdrawal due to insufficient clinical response | Study endpoint
Physician's Global Assessment of Disease Activity | Screening, Baseline, Week 1, Week 6, and Week 12
swollen joint count | Screening, Baseline, Week 1, Week 6, and Week 12
Adverse events | Baseline, Week 1, Week 6, and Week 12
Average rescue medication usage per day | Study endpoint
Short Form-36 Acute Health Survey | Baseline, Week 1, Week 6, and Week 12
tender joint count | Screening, Baseline, Week 1, Week 6, and Week 12
One-Week Severity of Dyspepsia Assessment | Baseline, Week 1, and Week 12
C-reactive protein | Screening, Baseline, Week 1, Week 6, and Week 12
laboratory tests | Screening, Baseline, Week 1, Week 6, and Week 12
vital signs | Screening, Baseline, Week 1, Week 6, and Week 12
physical examinations | Screening and Week 12
ACR-N | Study endpoint
Patient Treatment Satisfaction Scale | Week 1 and Week 6
Patient's assessment of arthritis pain (VAS) | Screening, Baseline, Week 1, Week 6, and Week 12
Health Assessment Questionnaire (HAQ) Disability Index | Screening, Baseline, Week 1, Week 6, and Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (52):
- United States (49):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, Glendale, Arizona
  - Pfizer Investigational Site, Mesa, Arizona
  - Pfizer Investigational Site, Paradise Valley, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Scottsdale, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Fullerton, California
  - Pfizer Investigational Site, Rancho Mirage, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Fort Lauderdale, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Jupiter, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Palm Harbor, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Zephyrhills, Florida
  - Pfizer Investigational Site, Idaho Falls, Idaho
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Springfield, Illinois
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Frederick, Maryland
  - Pfizer Investigational Site, Greenbelt, Maryland
  - Pfizer Investigational Site, Lansing, Michigan
  - Pfizer Investigational Site, Jackson, Mississippi
  - Pfizer Investigational Site, Marlton, New Jersey
  - Pfizer Investigational Site, Passaic, New Jersey
  - Pfizer Investigational Site, Teaneck, New Jersey
  - Pfizer Investigational Site, Brooklyn, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Allentown, Pennsylvania
  - Pfizer Investigational Site, Duncansville, Pennsylvania
  - Pfizer Investigational Site, Erie, Pennsylvania
  - Pfizer Investigational Site, Johnstown, Pennsylvania
  - Pfizer Investigational Site, Mechanicsburg, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Philadephia, Pennsylvania
  - Pfizer Investigational Site, Providence, Rhode Island
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, El Paso, Texas
  - Pfizer Investigational Site, Fort Worth, Texas
  - Pfizer Investigational Site, Plano, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Arlington, Virginia
  - Pfizer Investigational Site, Seattle, Washington
- Canada (3):
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Windsor, Ontario
  - Pfizer Investigational Site, Saskatoon, Saskatchewan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3471018&StudyName=Efficacy%20and%20Safety%20of%20valdecoxib%20and%20Naproxen%20in%20Treating%20the%20Signs%20and%20Symptoms%20of%20Rheumatoid%20Arthritis%20%28RA%29%20in%20a%20Severe%20Rheumat